CLINICAL TRIAL: NCT04309487
Title: Diagnostic Accuracy of ShuntCheck Compared With Radionuclide Shunt Patency Test to Detect Shunt Flow Obstruction in Patients With Normal Pressure Hydrocephalus - A Cross-sectional Analytic Study
Brief Title: Diagnostic Accuracy of ShuntCheck Compared to Radionuclide Shunt: Patency in Patients With Normal Pressure Hydrocephalus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Collaborators: NeuroDx Development (Industry)
Responsible Party: Principal Investigator, Naomi Abel, Assistant Professor, College of Medicine Neurosurgery, University of South Florida
Other Study IDs: Pro00041345
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Hydrocephalus, Normal Pressure
Keywords: Asymptomatic Normal Pressure Hydrocephalus; Ventriculoperitoneal Shunt
MeSH Terms: conditions — Hydrocephalus, Normal Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ShuntCheck: Participants will be administered the ShuntCheck diagnostic test.
  Interventions: Diagnostic Test: ShuntCheck

INTERVENTIONS:
Diagnostic Test: ShuntCheck — The intervention is an FDA-cleared device utilizing a transcutaneous thermal convection to analyze shunt flow.

SUMMARY:
The purpose of this study is to assess the diagnostic accuracy of ShuntCheck compared with radionuclide shunt patency testing (SPS) to detect CSF shunt flow of NPH patients with suspected shunt obstruction.

DETAILED DESCRIPTION:
The purpose of this study is to assess the diagnostic accuracy of ShuntCheck compared with radionuclide shunt patency testing (SPS) to detect CSF shunt flow of NPH patients with suspected shunt obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 40 yo or older and have a VP shunt placed for NPH and are suspected of shunt obstruction.
* Capable of providing valid signed informed consent, or has a legal guardian, health care agent, or surrogate decision maker (according to local statutes, and collectively referred to as "surrogates" in this protocol) capable of providing valid, signed informed consent

Exclusion Criteria:

* Presence of multiple shunts, or presence of more than one distal shunt catheter (regardless of function) crossing the clavicle ipsilateral to the shunt with suspected obstruction;
* ShuntCheck test would interfere with standard patient care, or emergency shunt surgery that cannot be delayed is indicated;
* Presence of an interfering open wound or edema over any portion of the VP shunt.

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of NPH hydrocephalus research subjects who have a VP shunt with a single ventricular catheter implanted for adult hydrocephalus are suspected of shunt obstruction and are scheduled for a radionuclide SPS.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-01-24 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of ShuntCheck compared to radionuclide shunt patency study | 15 minutes
Negative Predictive Value of ShuntCheck compared to radionuclide shunt patency study | 60 Minutes

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Abel, MD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida Department of Neurological Surgery and Brain Repair, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No
At present there is no plan to share any individual participant data.